CLINICAL TRIAL: NCT05025228
Title: Analgesic Effect of Paracetamol in Patients With Femur Fracture: is Intravenous Better Than Oral?
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Prot. 36041/19 ID: 2727
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2020-06

CONDITIONS: Femur Fracture
Keywords: Femur Fracture; Pain; Paracetamol; Emergency Department
MeSH Terms: conditions — Femoral Fractures; Pain; Emergencies | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Paracetamol IV: Patients with femur fracture that received an initial analgesic treatment with paracetamol intravenously (IV).
  Interventions: Drug: Paracetamol
- Paracetamol OR: Patients with femur fracture that received an initial analgesic treatment with paracetamol orally (OR).
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Paracetamol given orally or intravenously
  Other Names: Acetaminophen; N-acetyl-para-aminophenol

SUMMARY:
The purpose of this study is to monitor severe pain for femur fracture after treatment with paracetamol IV or OR.

DETAILED DESCRIPTION:
The investigators enrolled 170 consecutive patients with femur fracture and severe pain. The patients received an initial analgesic treatment with paracetamol orally (OR) or intravenously (IV). The primary outcome was the reduction of pain of 1 point at visual analogue scale for pain (VAS) after the 1 st hour of treatment (T1). Secondary endpoints included the reduction of pain of at least 2 points on the VAS scale at the 4 th hour (T4), the need of rescue therapy and the number of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients admitted to the ED of Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
* Femur Fracture
* Patients who signed the informed consent
* Able to take analgesic therapy both orally (OR) and intravenously (IV)
* Able to define pain by VAS

Exclusion Criteria:

* Age <18 years
* Allergy to paracetamol
* Unable to take analgesic therapy both orally (OR) and intravenously (IV)
* Unable to define pain by VAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with femur fracture admitted to the ED of Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pain change of 1 point at visual analogue scale for pain (VAS) after the 1 st hour of treatment (T1). | Baseline and 1 hour
  The Visual Analogue Scale for Pain (VAS) is a validated self-reported instrument that identifies pain from 0 to 10 (with 0 = no pain and 10 = maximum pain intensity)

SECONDARY OUTCOMES:
Pain change of at least 2 points on the VAS scale at the 4 th hour (T4) | Baseline and 4 hours
  identifies pain from 0 to 10 (with 0 = no pain and 10 = maximum pain intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franceschi, Study Director — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results of the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available immediately and ending 3 years after the publication of the study.
Access Criteria: Proposals should be directed to francesco.franceschi@policlinicogemelli.it. To gain access, requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Dizdarevic A, Farah F, Ding J, Shah S, Bryan A, Kahn M, Kaye AD, Gritsenko K. A Comprehensive Review of Analgesia and Pain Modalities in Hip Fracture Pathogenesis. Curr Pain Headache Rep. 2019 Aug 6;23(10):72. doi: 10.1007/s11916-019-0814-9. PMID 31388846
- [Background] Gangavalli AK, Nwachuku CO. Management of Distal Femur Fractures in Adults: An Overview of Options. Orthop Clin North Am. 2016 Jan;47(1):85-96. doi: 10.1016/j.ocl.2015.08.011. PMID 26614924
- [Background] Glinkowski W, Narloch J, Krasuski K, Sliwczynski A. The Increase of Osteoporotic Hip Fractures and Associated One-Year Mortality in Poland: 2008-2015. J Clin Med. 2019 Sep 18;8(9):1487. doi: 10.3390/jcm8091487. PMID 31540458
- [Background] Soffin EM, Gibbons MM, Wick EC, Kates SL, Cannesson M, Scott MJ, Grant MC, Ko SS, Wu CL. Evidence Review Conducted for the Agency for Healthcare Research and Quality Safety Program for Improving Surgical Care and Recovery: Focus on Anesthesiology for Hip Fracture Surgery. Anesth Analg. 2019 Jun;128(6):1107-1117. doi: 10.1213/ANE.0000000000003925. PMID 31094775
- [Background] Fabi DW. Multimodal Analgesia in the Hip Fracture Patient. J Orthop Trauma. 2016 May;30 Suppl 1:S6-S11. doi: 10.1097/BOT.0000000000000561. PMID 27101321
- [Background] Elsoe R, Ceccotti AA, Larsen P. Population-based epidemiology and incidence of distal femur fractures. Int Orthop. 2018 Jan;42(1):191-196. doi: 10.1007/s00264-017-3665-1. Epub 2017 Nov 7. PMID 29116356
- [Background] Bonnin MP, Neto CC, Aitsiselmi T, Murphy CG, Bossard N, Roche S. Increased incidence of femoral fractures in small femurs and women undergoing uncemented total hip arthroplasty - why? Bone Joint J. 2015 Jun;97-B(6):741-8. doi: 10.1302/0301-620X.97B6.35022. PMID 26033052
- [Background] Lim SJ, Yeo I, Yoon PW, Yoo JJ, Rhyu KH, Han SB, Lee WS, Song JH, Min BW, Park YS. Incidence, risk factors, and fracture healing of atypical femoral fractures: a multicenter case-control study. Osteoporos Int. 2018 Nov;29(11):2427-2435. doi: 10.1007/s00198-018-4640-4. Epub 2018 Jul 23. PMID 30039251
- [Background] Mattisson L, Bojan A, Enocson A. Epidemiology, treatment and mortality of trochanteric and subtrochanteric hip fractures: data from the Swedish fracture register. BMC Musculoskelet Disord. 2018 Oct 12;19(1):369. doi: 10.1186/s12891-018-2276-3. PMID 30314495
- [Background] Roder F, Schwab M, Aleker T, Morike K, Thon KP, Klotz U. Proximal femur fracture in older patients--rehabilitation and clinical outcome. Age Ageing. 2003 Jan;32(1):74-80. doi: 10.1093/ageing/32.1.74. PMID 12540352
- [Background] Larsen P, Ceccotti AA, Elsoe R. High mortality following distal femur fractures: a cohort study including three hundred and two distal femur fractures. Int Orthop. 2020 Jan;44(1):173-177. doi: 10.1007/s00264-019-04343-9. Epub 2019 May 12. PMID 31081515
- [Background] Rowlands M, Walt GV, Bradley J, Mannings A, Armstrong S, Bedforth N, Moppett IK, Sahota O. Femoral Nerve Block Intervention in Neck of Femur Fracture (FINOF): a randomised controlled trial. BMJ Open. 2018 Apr 10;8(4):e019650. doi: 10.1136/bmjopen-2017-019650. PMID 29643155
- [Background] Uysal AI, Altiparmak B, Yasar E, Turan M, Canbek U, Yilmaz N, Gumus Demirbilek S. The effects of early femoral nerve block intervention on preoperative pain management and incidence of postoperative delirium geriatric patients undergoing trochanteric femur fracture surgery: A randomized controlled trial. Ulus Travma Acil Cerrahi Derg. 2020 Jan;26(1):109-114. doi: 10.14744/tjtes.2019.78002. PMID 31942744
- [Background] Oc Y, Varol A, Yazar EA, Ak S, Akpolat AO, Kilinc BE. Treatment strategy for elderly patients with the isolated greater trochanteric fracture. SAGE Open Med. 2020 Oct 7;8:2050312120964138. doi: 10.1177/2050312120964138. eCollection 2020. PMID 33101681
- [Background] Li L, Bennett-Brown K, Morgan C, Dattani R. Hip fractures. Br J Hosp Med (Lond). 2020 Aug 2;81(8):1-10. doi: 10.12968/hmed.2020.0215. PMID 32845763
- [Background] Makkar JK, Jain K, Kuberan A, Balasubramanian M, Bhatia N, Singh PM. Pre-emptive multimodal analgesic regimen reduces post-operative epidural demand boluses in traumatic shaft of femur fracture - A randomised controlled trial. Indian J Anaesth. 2019 Nov;63(11):895-899. doi: 10.4103/ija.IJA_363_19. Epub 2019 Nov 8. PMID 31772397
- [Background] Chuang PY, Shen SH, Yang TY, Huang TW, Huang KC. Non-steroidal anti-inflammatory drugs and the risk of a second hip fracture: a propensity-score matching study. BMC Musculoskelet Disord. 2016 May 4;17:201. doi: 10.1186/s12891-016-1047-2. PMID 27141945
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Franceschi F, Marsiliani D, Alesi A, Mancini MG, Ojetti V, Candelli M, Gabrielli M, D'Aurizio G, Gilardi E, Adducci E, Proietti R, Buccelletti F. A simplified way for the urgent treatment of somatic pain in patients admitted to the emergency room: the SUPER algorithm. Intern Emerg Med. 2015 Dec;10(8):985-92. doi: 10.1007/s11739-015-1304-7. Epub 2015 Sep 4. PMID 26341218
- [Background] Di Filippo A, Magherini M, Ruggiano P, Ciardullo A, Falsini S. Postoperative analgesia in patients older than 75 years undergoing intervention for per-trochanteric hip fracture: a single centre retrospective cohort study. Aging Clin Exp Res. 2015 Jun;27(3):281-5. doi: 10.1007/s40520-014-0272-5. Epub 2014 Sep 17. PMID 25227548
- [Background] Aprato A, Bechis M, Buzzone M, Bistolfi A, Daghino W, Masse A. No rest for elderly femur fracture patients: early surgery and early ambulation decrease mortality. J Orthop Traumatol. 2020 Aug 30;21(1):12. doi: 10.1186/s10195-020-00550-y. PMID 32862297
- [Background] Mubark I, Abouelela A, Genena A, Al Ghunimat A, Sarhan I, Ashwood N. Mortality Following Distal Femur Fractures Versus Proximal Femur Fractures in Elderly Population: The Impact of Best Practice Tariff. Cureus. 2020 Sep 30;12(9):e10744. doi: 10.7759/cureus.10744. PMID 33150119
- [Background] Kanis JA, Oden A, McCloskey EV, Johansson H, Wahl DA, Cooper C; IOF Working Group on Epidemiology and Quality of Life. A systematic review of hip fracture incidence and probability of fracture worldwide. Osteoporos Int. 2012 Sep;23(9):2239-56. doi: 10.1007/s00198-012-1964-3. Epub 2012 Mar 15. PMID 22419370
- [Background] Piscitelli P, Neglia C, Feola M, Rizzo E, Argentiero A, Ascolese M, Rivezzi M, Rao C, Miani A, Distante A, Esposito S, Iolascon G, Tarantino U. Updated incidence and costs of hip fractures in elderly Italian population. Aging Clin Exp Res. 2020 Dec;32(12):2587-2593. doi: 10.1007/s40520-020-01497-0. Epub 2020 Feb 13. PMID 32056151
- [Background] Guzon-Illescas O, Perez Fernandez E, Crespi Villarias N, Quiros Donate FJ, Pena M, Alonso-Blas C, Garcia-Vadillo A, Mazzucchelli R. Mortality after osteoporotic hip fracture: incidence, trends, and associated factors. J Orthop Surg Res. 2019 Jul 4;14(1):203. doi: 10.1186/s13018-019-1226-6. PMID 31272470
- [Background] Peeters CM, Visser E, Van de Ree CL, Gosens T, Den Oudsten BL, De Vries J. Quality of life after hip fracture in the elderly: A systematic literature review. Injury. 2016 Jul;47(7):1369-82. doi: 10.1016/j.injury.2016.04.018. Epub 2016 Apr 23. PMID 27178770
- [Background] Mian P, Allegaert K, Spriet I, Tibboel D, Petrovic M. Paracetamol in Older People: Towards Evidence-Based Dosing? Drugs Aging. 2018 Jul;35(7):603-624. doi: 10.1007/s40266-018-0559-x. PMID 29916138
- [Background] Gazelka HM, Leal JC, Lapid MI, Rummans TA. Opioids in Older Adults: Indications, Prescribing, Complications, and Alternative Therapies for Primary Care. Mayo Clin Proc. 2020 Apr;95(4):793-800. doi: 10.1016/j.mayocp.2020.02.002. PMID 32247352
- [Background] Gemmati D, Varani K, Bramanti B, Piva R, Bonaccorsi G, Trentini A, Manfrinato MC, Tisato V, Care A, Bellini T. "Bridging the Gap" Everything that Could Have Been Avoided If We Had Applied Gender Medicine, Pharmacogenetics and Personalized Medicine in the Gender-Omics and Sex-Omics Era. Int J Mol Sci. 2019 Dec 31;21(1):296. doi: 10.3390/ijms21010296. PMID 31906252
- [Background] Di Sanzo M, Cipolloni L, Borro M, La Russa R, Santurro A, Scopetti M, Simmaco M, Frati P. Clinical Applications of Personalized Medicine: A New Paradigm and Challenge. Curr Pharm Biotechnol. 2017;18(3):194-203. doi: 10.2174/1389201018666170224105600. PMID 28240172
- [Result] Dixon J, Ashton F, Baker P, Charlton K, Bates C, Eardley W. Assessment and Early Management of Pain in Hip Fractures: The Impact of Paracetamol. Geriatr Orthop Surg Rehabil. 2018 Oct 25;9:2151459318806443. doi: 10.1177/2151459318806443. eCollection 2018. PMID 30377550